CLINICAL TRIAL: NCT03736720
Title: Phase 2 Single-Arm Study of Nanoliposomal Irinotecan With Fluorouracil and Leucovorin in Refractory Advanced High Grade Neuroendocrine Cancer of GI, Unknown or Pancreatic Origin
Brief Title: Liposomal Irinotecan, Fluorouracil and Leucovorin in Treating Patients With Refractory Advanced High Grade Neuroendocrine Cancer of Gastrointestinal, Unknown, or Pancreatic Origin
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: i 64518; NCI-2018-02122 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); i 64518 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2018-11-05; First posted 2018-11-09 (Actual); Results first posted 2023-12-19 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Locally Advanced Digestive System Neuroendocrine Carcinoma; Locally Advanced Pancreatic Neuroendocrine Carcinoma; Metastatic Digestive System Neuroendocrine Carcinoma; Metastatic Pancreatic Neuroendocrine Carcinoma; Refractory Digestive System Neuroendocrine Carcinoma; Refractory Pancreatic Neuroendocrine Carcinoma; Unresectable Digestive System Neuroendocrine Carcinoma; Unresectable Pancreatic Neuroendocrine Carcinoma
MeSH Terms: conditions — Somatostatinoma | interventions — Fluorouracil; dehydroftorafur; Leucovorin; irinotecan sucrosofate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (liposomal irinotecan, leucovorin, fluorouracil) (Experimental): Patients receive liposomal irinotecan IV over 90 minutes, leucovorin IV over 30 minutes, and fluorouracil IV over 46 hours on days 1 and 15. Courses repeat every 28 days for in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fluorouracil; Drug: Leucovorin; Drug: Liposomal Irinotecan; Procedure: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Leucovorin — Given IV
  Other Names: Folinic acid
Drug: Liposomal Irinotecan — Given IV
  Other Names: Irinotecan Liposome; MM-398; nal-IRI; Nanoliposomal Irinotecan; Nanoparticle Liposome Formulation of Irinotecan; Onivyde; PEP02
Procedure: Quality-of-Life Assessment — Correlative studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies how well liposomal irinotecan, leucovorin, and fluorouracil work in treating patients with high grade neuroendocrine cancer of gastrointestinal, unknown, or pancreatic origin that does not respond to treatment and has spread to other places in the body. Lliposomal irinotecan may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as fluorouracil and leucovorin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving liposomal irinotecan, leucovorin and fluorouracil may work better in treating patients with neuroendocrine cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rate liposomal irinotecan (nanoliposomal irinotecan [Nal-IRI]) + fluorouracil (5FU) and leucovorin in patients with refractory advanced high grade neuroendocrine cancer of gastrointestinal (GI), unknown or pancreatic origin.

SECONDARY OBJECTIVES:

I. To determine overall survival, progression-free survival, time to treatment failure, safety, clinical response and, quality of life (QOL) changes resulting from the combination treatment of nanoliposomal irinotecan (Nal-IRI) + fluorouracil (5FU) and leucovorin.

EXPLORATORY OBJECTIVES:

I. Genetic profiling for mutations will be conducted on all pre-study tumor samples and compared to changes in immune response.

OUTLINE:

Patients receive liposomal irinotecan intravenously (IV) over 90 minutes, leucovorin IV over 30 minutes, and fluorouracil IV over 46 hours on days 1 and 15. Courses repeat every 28 days for in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days, then every 2 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a locally advanced and unresectable or metastatic gastroenteropancreatic neuroendocrine carcinoma of the gastrointestinal (GI) tract, pancreas, or of other known or unknown primary site where 5FU based therapy would be considered reasonable by the treated MD, lung primary is excluded. Patients may have either progressed on therapy or within 6 months of completing therapy, or be intolerant of therapy to be considered eligible.
* Participant must have tissue available for central pathology review and, must have pathologically/histologically confirmed high grade neuro endocrine defined as Ki-67 proliferative index of 20-100% or, must have evidence of at least 10 mitotic figures per 10 high powered fields.
* Comprehensive Genomic Profiling will be performed on archival tissue available prior to enrollment. If no archival tissue is available, then patient must have fresh biopsy prior to treatment administration if clinically indicated.
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 - 2.
* Leukocytes >= 3,000/mm^3 .
* Absolute neutrophil count >= 1,500/mm^3.
* Hemoglobin >= 9 g/dL.
* Platelets >= 100,000/mm^3.
* Total bilirubin =< institutional upper limit of normal (ULN) or =< 1.5 x institutional ULN (if the patient has liver metastases.
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN or (=< 5 x institutional ULN if the patient has liver metastases).
* Serum creatinine =< 1.5 x institutional ULN or measured or calculated creatinine clearance by Cockcroft Gault Equation >= 50ml/min for subjects with creatinine levels > 1.5 x ULN.
* Have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria present.
* Participant must have a life expectancy of >= 12 weeks as determined clinically by the treating physician.
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

  * A female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
  * Women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception or to abstain from sexual intercourse for the duration of their participation in the study.
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Participants with known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
* Known hypersensitivity to any of the components of Nal-IRI, other liposomal products, fluoropyrimidines or leucovorin.
* Investigational therapy administered within 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is longer, prior to the first scheduled day of dosing in this study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or nursing female participants.
* Unwilling or unable to follow protocol requirements.
* Any condition which in the Investigator?s opinion deems the participant an unsuitable candidate to receive study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2024-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renuka Iyer, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Stony Brook Cancer Center, Stony Brook, New York

REFERENCES:
- [Derived] Abstracts Presented at the 13th Annual Multidisciplinary Neuroendocrine Tumor Medical Virtual Symposium of the North American Neuroendocrine Tumor Society, October 2-3, 2020. Pancreas. 2021 Mar 1;50(3):441-467. doi: 10.1097/MPA.0000000000001763. No abstract available. PMID 33835977

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Liposomal Irinotecan, Leucovorin, Fluorouracil)
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Liposomal Irinotecan, Leucovorin, Fluorouracil)
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 11
Number of Prior Chemotherapy Regimens [Count of Participants; unit: Participants] — The number of prior chemotherapy regimens for the current cancer diagnsosis.
  Participants
    No Prior Regimens | 0
    1 Prior Regimen | 7
    2 Prior Regimens | 3
    Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Description: Will be summarized using frequencies and relative frequencies; with the ORR (= CR+PR / N) estimated using an 80% confidence interval obtained using Jeffrey's prior method. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Within 6 months of treatment initiation
Population: 2 patients were not evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Liposomal Irinotecan, Leucovorin, Fluorouracil)
Number analyzed (Participants) | 9
Participants
  Objective Response (CR+PR) | 1
  No Objective Response (SD+PD) | 8
Statistical Analysis 1: Comparison: Treatment (Liposomal Irinotecan, Leucovorin, Fluorouracil); Test type: Other — No statistical test; Proportion = 0.091, 80% CI 2-sided [0.033 to 0.301] — Estimated using Jeffrey's prior method

2. Secondary Outcome: Overall Survival
Description: Will be summarized using standard Kaplan-Meier methods; where estimates of the median time will be obtained with 95% confidence intervals.
Time Frame: From first dosing of study treatment combination to time of death or imitation of a new therapy, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Liposomal Irinotecan, Leucovorin, Fluorouracil)
Number analyzed (Participants) | 11
months | 8.3 [2.3 to 18.2]

3. Secondary Outcome: Progression-free Survival Assessed by RECIST 1.1
Description: Will be summarized using standard Kaplan-Meier methods; where estimates of the median time will be obtained with 95% confidence intervals. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From first dosing of study treatment combination to disease progression, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Liposomal Irinotecan, Leucovorin, Fluorouracil)
Number analyzed (Participants) | 11
months | 3.9 [0.5 to 5.1]

4. Secondary Outcome: Time-to Treatment Failure
Description: Will be summarized using standard Kaplan-Meier methods; where estimates of the median time will be obtained with 90% confidence intervals.
Time Frame: From enrollment to discontinuation of treatment, assessed up to 3 years
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Liposomal Irinotecan, Leucovorin, Fluorouracil)
Number analyzed (Participants) | 11
months | 3.9 [1.7 to 4.4]

5. Secondary Outcome: Proportion of Patients Achieving an Objective Response Based on Prior Response to Platinum Etoposide
Description: The objective response rate (ORR) is as described in the primary analysis. Here it is reported in the subset of patients that received prior platinum etoposide therapy.
Time Frame: Up to 3 years
Population: Only 4 patients received prior platinum etoposide.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Liposomal Irinotecan, Leucovorin, Fluorouracil)
Number analyzed (Participants) | 4
Participants
  No Objective Response | 3
  Objective Response | 1

6. Secondary Outcome: Clinical Benefit Response
Description: Defined as either achievement of pronounced and sustained (>=4 weeks contiguous) improvement in pain intensity, analgesic consumption, or performance status, or a combination of these, without any worsening in any of the other factors, or stability in pain intensity, analgesic consumption, and performance status with pronounced and sustained (>= 4 weeks contiguous) weight gain. Will be treated as binary data and summarized using frequencies and relative frequencies. The clinical benefit response rate will be estimated using a 90% confidence interval obtained by Jeffrey?s prior method.
Time Frame: Up to 3 years
Population: The appropriate data to identify patient clinical benefit status (as defined above) was not adequately obtained (no available data) and analysis can not be conducted for this outcome measure.
Arm/Group | Treatment (Liposomal Irinotecan, Leucovorin, Fluorouracil)
Number analyzed (Participants) | 0

7. Secondary Outcome: Quality of Life (QOL) as Assessed by European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30)
Description: Will be treated as quantitative data and summarized by time-point using the mean and standard deviation. The QOL scores at each follow-up time may be compared with base-line levels using the paired t-test or sign test. The overall QoL rating ranges from 0 (poor) to 10 (good).
Time Frame: From treatment initiation until treatment completion/progression (up to 3 years).
Population: There are 11 patients that have QoL data at baseline (pre-treatment). There are only 8 patients with end of treatment QoL assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment (Liposomal Irinotecan, Leucovorin, Fluorouracil)
Number analyzed (Participants) | 11
units on a scale
  Pre Treatment QoL | 5.9 (1.4)
  End of Treatment QoL: number analyzed (Participants) | 8
  End of Treatment QoL | 5.5 (1.7)
Statistical Analysis 1: Comparison: Treatment (Liposomal Irinotecan, Leucovorin, Fluorouracil); Comparing the pre-treatment and end of treatment QoL scores; Test type: Superiority; p = 0.289, Sign test; two-sided test

8. Secondary Outcome: Incidence of Grade 3+ Treatment Related Adverse Events (TRAE)
Description: Toxicities and adverse events will be summarized by attribution and grade using frequencies and relative frequencies. High grade (3+) toxicity and adverse event rates may be estimated using 90% confidence intervals obtained by Jeffrey's prior method. Data Safety Monitoring Board (DSMB) monitoring will also occur periodically to ensure safety of study subjects.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Liposomal Irinotecan, Leucovorin, Fluorouracil)
Number analyzed (Participants) | 11
Participants
  No Grade 3+ TRAE | 4
  Grade 3+ TRAE | 7

ADVERSE EVENTS:
Time Frame: Adverse events were followed for up to 3 years following treatment initiation, with a median time of 182 days.
Arm/Group | Treatment (Liposomal Irinotecan, Leucovorin, Fluorouracil)
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 6/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Liposomal Irinotecan, Leucovorin, Fluorouracil) (N=11)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Other (Hepatobiliary disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Liposomal Irinotecan, Leucovorin, Fluorouracil) (N=11)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5)
Fatigue (General disorders) | 5 (5)
Sepsis (Infections and infestations) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Metabolism and nutrition disorders **Any AE - Maximum Grade Seen Hypokalemia Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Superior vena cava syndrome (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT03736720/Prot_SAP_000.pdf